CLINICAL TRIAL: NCT06329713
Title: The Effect of Changing the Programmed Auto Bolus Interval Time On Analgesic Quality of Labor Analgesia With Dural Puncture Epidural Technique: Double-Blind Randomised Controlled Study
Brief Title: Effect of Auto-Bolus Interval on Analgesic Quality During Labor Analgesia With Dural Puncture Epidural
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-03/11
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30-Min Interval (Active Comparator): The patients will be given 10 ml of a solution containing 0,1% of bupivacaine and 2 mcg/ml fentanyl through the epidural cathether. Level of sensory block will be tested by testing with ice from S2 dermatome cephally.
  Analgesia will be maintained by programmed intermittant epidural (PIE) boluses of 7,5 ml of 0,0625% of bupivacaine and 2 mcg/ml fentanyl every 30 minutes, starting 1 hour after the loading dose. In addition, patient controlled epidural analgesia (PCEA) will be programmed so that 8 ml of the same solution with a lock-time of 15 minutes may be administered. "Breakthrough pain" that requires even further analgesia will be treated with an epidural bolus of 10 ml of 0,1% bupivacain solution.
  Interventions: Procedure: Group I: 30 Min Interval Time
- 60-Min Interval (Active Comparator): The patients will be given 10 ml of a solution containing 0,1% of bupivacaine and 2 mcg/ml fentanyl through the epidural cathether. Level of sensory block will be tested by testing with ice from S2 dermatome cephally.
  Analgesia will be maintained by programmed intermittant epidural boluses of 15 ml of 0,0625% of bupivacaine and 2 mcg/ml fentanyl once in every hour, starting 1 hour after the loading dose. In addition, patient controlled epidural analgesia (PCEA) will be programmed so that 8 ml of the same solution with a lock-time of 15 minutes may be administered. "Breakthrough pain" that requires even further analgesia will be treated with an epidural bolus of 10 ml of 0,1% bupivacain solution.
  Interventions: Procedure: Group II: 60 Min Interval Time

INTERVENTIONS:
Procedure: Group I: 30 Min Interval Time — 10 ml of a solution containing 0,1% of bupivacaine and 2 mcg/ml fentanyl through the epidural cathether, maintained by programmed intermittant epidural (PIE) boluses of 7,5 ml of the same solution once in every 30 minutes, starting 1 hour after the loading dose. patient controlled epidural analgesia (PCEA) will be programmed so that 8 ml of the same solution with a lock-time of 15 minuts may be administered
  Arms: 30-Min Interval
Procedure: Group II: 60 Min Interval Time — 10 ml of a solution containing 0,1% of bupivacaine and 2 mcg/ml fentanyl through the epidural cathether, maintained by programmed intermittant epidural (PIE) boluses of 15 ml of the same solution once in every hour, starting 1 hour after the loading dose. patient controlled epidural analgesia (PCEA) will be programme
  Arms: 60-Min Interval

SUMMARY:
It is aimed in this study to compare the effect of changing the interval time for programmed auto boluses of local anaesthetics on the total anesthetic consumption and quality of labor analgesia with dural puncture epidural technique.

DETAILED DESCRIPTION:
This study will be conducted as a prospective randomized, controlled, double-blind trial following the approval of the ethical committee at Atatürk University Medical Faculty Hospital and after obtaining written consent from the participating patients. The study will include pregnant women aged 20 to 45 with American Society of Anesthesiologists (ASA) II classification, full-term, nulliparous and singleton pregnancies. Using a randomisation procedure, the participants will be allocated into two equal groups: Group I and Group II.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy nulliparous women
2. American Society of Anaesthesiology Score of II
3. During active labor
4. At weeks 37-42.
5. Singlet vertex presentation
6. Cervical dilation <5 cm at the request of labor analgesia
7. VAS score >40

Exclusion Criteria:

1. Age <20 or >45,
2. Morbid obesity
3. Presence of pregnancy-related comorbidities (e.g: gestational diebetes, gestational hypertension and preeclampsia)
4. History of drug abuse
5. Contrindication for neuraxial blocks
6. Conditions that increase the risk of need for cesarean section (e.g. placenta previa, uterus abnormalities or surgeries)
7. Diagnosed fetal abnormalities
8. Cases where dura gets punctured unintendedly with the epiduralneedle
9. Cases where flow of cerebrospinal fluid (CSF) is not observed after dural puncture
10. Cases where a cesarean section is performed at any stage of labor
11. Cases where labor is completed in 1 hour from the start of analgesia procedure.

Exclusion Criteria:

-

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference between total local anaesthetic consumption | 5 hours or before if the labor is completed
  The study will involve monitoring the patients starting 2 minutes after the initial epidural dose, every 2 minutes during the first 20 minutes. Monitoring will continue at the 30th minute, and once in every 90 minutes for 5 hours or until labor is completed.
  Total bupivacain consumption will be calculated as follows: PIEB + PCEA + boluses by the clinician. Bupivacain consumption per hour will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Dostbil, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Suzuki N, Koganemaru M, Onizuka S, Takasaki M. Dural puncture with a 26-gauge spinal needle affects spread of epidural anesthesia. Anesth Analg. 1996 May;82(5):1040-2. doi: 10.1097/00000539-199605000-00028. PMID 8610864
- [Background] Thomas JA, Pan PH, Harris LC, Owen MD, D'Angelo R. Dural puncture with a 27-gauge Whitacre needle as part of a combined spinal-epidural technique does not improve labor epidural catheter function. Anesthesiology. 2005 Nov;103(5):1046-51. doi: 10.1097/00000542-200511000-00019. PMID 16249679
- [Background] Wilson SH, Wolf BJ, Bingham K, Scotland QS, Fox JM, Woltz EM, Hebbar L. Labor Analgesia Onset With Dural Puncture Epidural Versus Traditional Epidural Using a 26-Gauge Whitacre Needle and 0.125% Bupivacaine Bolus: A Randomized Clinical Trial. Anesth Analg. 2018 Feb;126(2):545-551. doi: 10.1213/ANE.0000000000002129. PMID 28622178
- [Background] Kaddoum R, Motlani F, Kaddoum RN, Srirajakalidindi A, Gupta D, Soskin V. Accidental dural puncture, postdural puncture headache, intrathecal catheters, and epidural blood patch: revisiting the old nemesis. J Anesth. 2014 Aug;28(4):628-30. doi: 10.1007/s00540-013-1761-y. Epub 2013 Dec 18. PMID 24347033